CLINICAL TRIAL: NCT02238626
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, 6-month Trial Followed by an Open-label Extension to Evaluate the Safety, Tolerability and Clinical Endpoint Responsiveness of Ibudilast (MN-166) in Subjects With (ALS)
Brief Title: Ibudilast (MN-166) in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Acronym: IBU-ALS-1201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediciNova (Industry)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MN-166-ALS-1201
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; pharmacotherapy; intervention; prospective; safety endpoint; preliminary efficacy; ibudilast
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Sugars; Tablets; ibudilast; Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (for MN-166) (Placebo Comparator): Sugar pill manufactured for MN-166 10 mg tablets plus 50 mg riluzole by mouth twice daily for 6 months.
  Interventions: Drug: Placebo (for MN-166); Drug: riluzole
- MN-166 (Experimental): MN-166 10 mg tablets (up to 60 mg/day) by mouth 2-3 times a day plus 50 mg riluzole 2 times a day by mouth for 6 months.
  Interventions: Drug: MN-166; Drug: riluzole

INTERVENTIONS:
Drug: Placebo (for MN-166)
  Other Names: Sugar pill manufactured to mimic MN-166 10 mg tablet
  Arms: Placebo (for MN-166)
Drug: MN-166
  Other Names: ibudilast
  Arms: MN-166
Drug: riluzole — Patient is given 50 mg riluzole twice daily.
  Other Names: Rilutek

SUMMARY:
This is a single center, randomized, double-blind, placebo-controlled, 6-month study designed to evaluate the safety, tolerability and clinical responsiveness of MN-166/ibudilast (60 mg/day) when administered as an adjunct to riluzole (100 mg/day) in 60 subjects with ALS.

This study will consist of two treatment arms, MN-166 and matching placebo. Randomization will occur in a 2:1 ratio (MN- 166: placebo).

Duration of Treatment: Screening Phase: up to 3 months; Double-blind Phase: 6 months; Open-label Phase 6 months (for placebo subjects only); Follow-up Phase: 2 weeks after last dose.

During treatment phase, subjects return to the clinic at Months 3 and 6 and will be telephoned by staff at Months 1,2,4, and 5 to collect information about side effects and new or concomitant medications.

All subjects (subjects who complete the Double-blind Phase and subjects who complete the Open-label Phase) or prematurely discontinue will return for a follow-up visit approximately 2 weeks after the last dose of study drug to assess adverse event status and to document concomitant medications.

Safety will be assessed by monitoring and recording all treatment-emergent adverse events (TEAEs) including serious adverse events (SAEs) and discontinuations due to TEAEs. Additional assessments will include regular monitoring of hematology, blood chemistry, and urine values, regular measurement of vital signs, ECGs, medical history, physical and neurological examinations.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained and willing and able to comply with the protocol in the opinion of the Investigator.
* Male or female subjects ages ≥ 18 to 80 years, inclusive
* Diagnosis of familial or sporadic ALS as defined by the El Escorial-Revised (2000) research diagnostic criteria for ALS [Clinically Definite, Clinically Probable, Probable-Laboratory-Supported]
* Diagnosis of ALS with onset of less than or equal to 5 years from first clinical weakness
* Slow vital capacity ≥ 60% of predicted within 1 month prior to Treatment Day 1
* Currently on a stable dose of riluzole for at least 30 days prior to initiation of study drug. Subjects not currently taking riluzole will be started on 50 mg qd for the first 7 days followed by 50 mg bid for the following 21 days prior to screening. Patients may be screened during this time period but not started on study drug until they are on a stable dose of riluzole.
* All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing). Females of childbearing potential must use an effective method of contraception throughout the entire study period and for 30 days after study drug discontinuation.
* Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
* Males should practice contraception as follows: condom use and contraception by female partner.
* Able to swallow study medication capsules.
* Subject is willing and able to comply with the protocol assessments and visits, in the opinion of the study nurse/coordinator and the Investigator.
* Has no known allergies to the study drug or its excipients.
* Has received 23-valent pneumococcal vaccine within 4 years prior to starting clinical trial.

Exclusion Criteria:

* Use of tracheostomy, tracheostomy invasive mechanical ventilation [TIMV].
* Greater than 3% predicted loss in post-diagnosis vital capacity per month or a greater than 1 unit loss in post diagnosis ALSFRS-R total score per month [ exclusive of loss due to beginning use of assistive devices]
* Confirmed hepatic insufficiency or abnormal liver function (AST and/or ALT greater than 3 times the upper limit of the normal range)
* Renal insufficiency as defined by a serum creatinine greater than 1.5 times the upper limit of normal range
* Currently has a clinically significant psychiatric disorder or dementia which would preclude evaluation of symptoms.
* Has a clinically significant medical condition (other than ALS) including the following: neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological disorder, or central nervous system infection that would pose a risk to the subject if they were to participate in the study or that might confound the results of the study.
* History of malignancy < 5 years prior to signing the informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* ECG finding of QTcB prolongation > 450 ms for males and > 470 ms for females at screening
* History of HIV (human immunodeficiency virus), clinically significant chronic hepatitis, or other active infection
* Subject has a history of stomach or intestinal surgery or any other condition that could interfere with or is judged by the Investigator to interfere with absorption, distribution, metabolism, or excretion of study drug.
* Subject has a history of alcohol or substance abuse (DSM-IV-TR criteria) within 3 months prior to screening or alcohol or substance dependence (DSM-IV-TR criteria) within 12 months prior to screening.
* Subject has poor peripheral venous access that will limit the ability to draw blood as judged by the Investigator.
* Currently participating, or has participated in, a study with an investigational or marketed compound or device within 3 months prior to signing the informed consent.
* Unable to cooperate with any study procedures, unlikely to adhere to the study procedures and keep appointments, in the opinion of the Investigator.

Advanced ALS group will follow the same inclusion/exclusion as the early ALS subjects with the exception of the following:

Inclusion criteria:

* Diagnosis of ALS with onset of ≤10 years from first clinical weakness
* On Non-invasive ventilator with Non-invasive pressure [P-NIV] or volume [V-NIV] cycled ventilation stable use for ≥ 4 hours daily for 1 month prior to Treatment Day.
* Slow vital capacity ≥ 20% of predicted (Knudsen 1983) within 1 month prior to Treatment Day 1
* Able to swallow study medication capsules or have gastrostomy tube access for delivery of contents of medication capsule.

Exclusion criteria:

* Use of tracheostomy, tracheostomy invasive mechanical ventilation [TIMV].
* No rate of progression exclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin R Brooks, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Healthcare System, Dept. of Neurology, Charlotte, North Carolina, United States

REFERENCES:
- See also: Please call 1-844-CMC-ALS1 (1-844-262-2571) toll free for information on this trial. — http://carolinashealthcare.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (for MN-166) (Early ALS Cohort): Sugar pill manufactured for MN-166 10 mg tablets plus 50 mg riluzole by mouth twice daily for 6 months.
  Placebo (for MN-166)
  riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS onset is 5 years or less.
- MN-166 (Early ALS Cohort): MN-166 10 mg tablets (up to 60 mg/day) by mouth 2-3 times a day plus 50 mg riluzole 2 times a day by mouth for 6 months.
  MN-166
  riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS onset is 5 years or less.
- Placebo (Advanced ALS Cohort): Sugar pill manufactured for MN-166 10 mg tablets plus 50 mg riluzole by mouth twice daily for 6 months.
  Placebo (for MN-166)
  riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS onset more than 5 years, but less than 10 years.
- MN-166 (Advanced ALS Cohort): MN-166 10 mg tablets (up to 60 mg/day) by mouth 2-3 times a day plus 50 mg riluzole 2 times a day by mouth for 6 months.
  MN-166
  riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS onset is less than 10 years, but more than 5 years.
Period: Overall Study
Arm/Group | Placebo (for MN-166) (Early ALS Cohort) | MN-166 (Early ALS Cohort) | Placebo (Advanced ALS Cohort) | MN-166 (Advanced ALS Cohort)
Started | 17 | 34 | 8 | 11
Completed | 12 | 20 | 5 | 4
Not Completed | 5 | 14 | 3 | 7
Not completed — Adverse Event | 3 | 5 | 0 | 3
Not completed — Lost to Follow-up | 2 | 4 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Other | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Early ALS Cohort: Patient ALS symptom onset 5 years or less before screening. Advanced ALS Cohort: Patient ALS symptom onset between 5 and 10 years before screening.
Groups:
- Placebo (for MN-166) (Early ALS Cohort): Sugar pill manufactured for MN-166 10 mg tablets plus 50 mg riluzole by mouth twice daily for 6 months.
  Placebo (for MN-166)
  riluzole: Patient is given 50 mg riluzole twice daily.
- MN-166 (Early ALS Cohort): MN-166 10 mg tablets (up to 60 mg/day) by mouth 2-3 times a day plus 50 mg riluzole 2 times a day by mouth for 6 months.
  MN-166
  riluzole: Patient is given 50 mg riluzole twice daily.
- Placebo (for MN-166) (Advanced ALS Cohort): Sugar pill manufactured for MN-166 10 mg tablets plus 50 mg riluzole by mouth twice daily for 6 months.
  Placebo (for MN-166) riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS symptom onset between 5 and 10 years of Screening.
- MN-166 (Advanced ALS Cohort): MN-166 10 mg tablets (up to 60 mg/day) by mouth 2-3 times a day plus 50 mg riluzole 2 times a day by mouth for 6 months.
  MN-166 riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS symptom onset between 5 and 10 years before screening.
- Total: Total of all reporting groups
Arm/Group | Placebo (for MN-166) (Early ALS Cohort) | MN-166 (Early ALS Cohort) | Placebo (for MN-166) (Advanced ALS Cohort) | MN-166 (Advanced ALS Cohort) | Total
Number analyzed (Participants) | 17 | 34 | 8 | 11 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (9.8) | 60.4 (10.9) | 56.9 (7.4) | 61.6 (8.1) | 58.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 2 | 5 | 23
  Male | 12 | 23 | 6 | 6 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 34 | 8 | 11 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 0 | 5
  White | 15 | 31 | 6 | 11 | 63
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 34 | 8 | 11 | 70

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of MN-166 60 mg/d Versus Placebo When Administered With Riluzole in Subjects With ALS
Description: Safety will be assessed by monitoring and recording all treatment-emergent adverse events (TEAEs) including serious adverse events (SAEs) and discontinuations due to TEAEs and Additional assessments will include regular monitoring of hematology, blood chemistry, and urine values, regular measurement of vital signs, ECGs, medical history, physical and neurological examinations.
Time Frame: 6 months
Population: Safety analysis population included all randomized subjects who received at least one dose of study drug and had at least one post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (for MN-166) (Early ALS Cohort): Sugar pill manufactured for MN-166 10 mg tablets plus 50 mg riluzole by mouth twice daily for 6 months.
  Placebo (for MN-166)
  riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS onset within 5 years.
- MN-166: MN-166 10 mg tablets (up to 60 mg/day) by mouth 2-3 times a day plus 50 mg riluzole 2 times a day by mouth for 6 months.
  MN-166
  riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS onset within 5 years.
- Placebo (for MN-166) (Advanced ALS Cohort): Sugar pill manufactured for MN-166 10 mg tablets plus 50 mg riluzole by mouth twice daily for 6 months.
  Placebo (for MN-166)
  riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS symptom onset between 5 and 10 years before Screening.
Arm/Group | Placebo (for MN-166) (Early ALS Cohort) | MN-166 | Placebo (for MN-166) (Advanced ALS Cohort) | MN-166 (Advanced ALS Cohort)
Number analyzed (Participants) | 17 | 34 | 8 | 11
Participants | 17 | 34 | 8 | 11

2. Secondary Outcome: Mean Change in Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised Total Score From Baseline to Month 6
Description: Functional activity as assessed by the Amyotrophic Lateral Sclerosis Functional Rating Scale-revised from baseline visit to Month 6. The best possible score is 48; the worst possible score is 0. Typically, ALS scores decline. In this outcome, the change in score will be a negative value, e.g., -4, -8, etc. The higher negative value indicates greater decline in functional activity (change in score -8 is worse than change in score -4).
Time Frame: 6 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo (for MN-166) (Early ALS Cohort): Sugar pill manufactured for MN-166 10 mg tablets plus 50 mg riluzole by mouth twice daily for 6 months.
  Placebo (for MN-166)
  riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS symptom onset within 5 years of Screening.
- MN-166 (Early ALS Cohort): MN-166 10 mg tablets (up to 60 mg/day) by mouth 2-3 times a day plus 50 mg riluzole 2 times a day by mouth for 6 months.
  MN-166
  riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS symptom onset within 5 years of screening.
Arm/Group | Placebo (for MN-166) (Early ALS Cohort) | MN-166 (Early ALS Cohort) | Placebo (for MN-166) (Advanced ALS Cohort) | MN-166 (Advanced ALS Cohort)
Number analyzed (Participants) | 17 | 34 | 8 | 11
score on a scale | -3.8 (3.91) | -4.5 (5.1) | -2.2 (2.56) | -4.8 (4.92)

3. Secondary Outcome: Respiratory Function
Description: Change in respiratory function (breathing capacity) from baseline to Month 6, as measured by slow vital capacity, in which the patient breathes into a spirometer slowly until the lungs are cleared of air. SVC is measured in liters (L). The greater the mean change from baseline to 6 months, the worse the outcome. For example, -10 is worse than -6.
Time Frame: 6 months
Population: Subjects who completed Month 6 (double-blind treatment phase)
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Placebo (for MN-166) Early ALS Cohort: Sugar pill manufactured for MN-166 10 mg tablets plus 50 mg riluzole by mouth twice daily for 6 months.
  Placebo (for MN-166)
  riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS onset within 5 years of screening.
- MN-166 (Early ALS Cohort): MN-166 10 mg tablets (up to 60 mg/day) by mouth 2-3 times a day plus 50 mg riluzole 2 times a day by mouth for 6 months.
  MN-166
  riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS onset within 5 years of screening.
Arm/Group | Placebo (for MN-166) Early ALS Cohort | MN-166 (Early ALS Cohort) | Placebo (for MN-166) (Advanced ALS Cohort) | MN-166 (Advanced ALS Cohort)
Number analyzed (Participants) | 14 | 32 | 5 | 9
Liters | -6.1 (9.33) | -10.1 (9.89) | -12.2 (7.07) | -11.1 (18.73)

4. Secondary Outcome: Muscle Strength
Description: Muscle strength measured by manual muscle testing (MMT) and instrumented hand-held dynamometry. Maximum muscle strength is assessed by measuring the best of 2 handgrips represented as kilograms (kg). The greater the change from baseline to month 6, the worse off the subject is. For example, a change of -0.50 is worse than -0.40.
Time Frame: 6 months
Population: Subjects who completed Month 6 (double-blind treatment phase)
Measure: Mean (Standard Deviation); unit: weight (kg)
Groups:
- Placebo (for MN-166) (Early ALS Cohort): Sugar pill manufactured for MN-166 10 mg tablets plus 50 mg riluzole by mouth twice daily for 6 months.
  Placebo (for MN-166)
  riluzole: Patient is given 50 mg riluzole twice daily. Patient ALS onset within 5 years of screening.
Arm/Group | Placebo (for MN-166) (Early ALS Cohort) | MN-166 (Early ALS Cohort) | Placebo (for MN-166) (Advanced ALS Cohort) | MN-166 (Advanced ALS Cohort)
Number analyzed (Participants) | 14 | 32 | 5 | 8
weight (kg) | -3.9 (5.37) | -4.9 (5.50) | -1.3 (2.37) | -4.4 (3.63)

5. Secondary Outcome: Use of Non-invasive Ventilation
Description: Non-invasive ventilation (NIV) utilization measured by clinically indicated prescription for NIV intervention and time to clinically indicated prescription for NIV intervention in each group (for early ALS subjects only). This is intended to count the number of subjects who had to go on non-invasive ventilation, as prescribed by the Principal Investigator, during study participation.
Time Frame: 6 months
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (for MN-166) (Early ALS Cohort) | MN-166 (Early ALS Cohort)
Number analyzed (Participants) | 16 | 33
Participants | 6 | 10

6. Secondary Outcome: The Mean Change in Baseline to Month 6 in Quality of Life as Measured by the Amyotrophic Lateral Sclerosis Assessment Questionnaire - 5
Description: A patient self-reported questionnaire specifically designed to measure 5 areas of health: physical mobility, activities of daily living and independence, eating and drinking, communication, and emotional functioning. The ALSAQ-5 is brief and easy to complete questionnaire and has undergone rigorous testing for validity, reliability, and sensitivity to change and has been shown to be a robust tool for assessing ALS. The lowest possible score is 0 and the highest possible score is 20. The greater the mean decrease from baseline to Month 6, the group was considered worse off. For example, -2 is worse than -1. The greater the mean increase from baseline to Month 6, the group was considered improved. For example, 2 is better than 1.
Time Frame: 6 months
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo (for MN-166): Sugar pill manufactured for MN-166 10 mg tablets plus 50 mg riluzole by mouth twice daily for 6 months.
  Placebo (for MN-166)
  riluzole: Patient is given 50 mg riluzole twice daily.
- MN-166: MN-166 10 mg tablets (up to 60 mg/day) by mouth 2-3 times a day plus 50 mg riluzole 2 times a day by mouth for 6 months.
  MN-166
  riluzole: Patient is given 50 mg riluzole twice daily.
Arm/Group | Placebo (for MN-166) | MN-166 | Placebo (for MN-166) (Advanced ALS Cohort) | MN-166 (Advanced ALS Cohort)
Number analyzed (Participants) | 14 | 32 | 6 | 9
score on a scale | 2.1 (3.00) | 1.6 (2.77) | -0.70 (2.07) | 4.8 (3.56)

7. Secondary Outcome: Clinical Global Impression of Change (CGIC)
Description: A scale used to provide a global rating of illness severity, improvement, and response to treatment. It is a 3-item observer rating scale and uses a 7-point rating scale. The scale was rated relative to the previous standard of care visit prior to randomization for entry, i.e., -3 much much much worse, -2 much much worse, - 1 much worse, 0 no change, +1 much better, +2 much much better, +3 much, much, much better. Ratings were provided by the Investigator. The greater the mean decrease from baseline to Month 6, the group was considered worse off. For example, -2 is worse than -1. The greater the mean increase from baseline to Month 6, the group was considered improved. For example, 2 is better than 1.
Time Frame: 6 months
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo (for MN-166) (Early ALS Cohort) | MN-166 (Early ALS Cohort) | Placebo (for MN-166) (Advanced ALS Cohort) | MN-166 (Advanced ALS Cohort)
Number analyzed (Participants) | 14 | 32 | 6 | 9
score on a scale | -1.0 (0.78) | -1.4 (0.75) | -1.3 (0.52) | -1.6 (0.73)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline to end of double-blind treatment (6 months).
Arm/Group | Placebo (for MN-166) (Early ALS Cohort) | MN-166 (Early ALS Cohort) | Placebo (for MN-166) (Advanced ALS Cohort) | MN-166 (Advanced ALS Cohort)
All-Cause Mortality (participants affected / at risk) | 0/17 | 1/34 | 1/8 | 1/11
Serious Adverse Events (participants affected / at risk) | 1/17 | 5/34 | 2/8 | 3/11
Other Adverse Events (participants affected / at risk) | 17/17 | 34/34 | 8/8 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (for MN-166) (Early ALS Cohort) (N=17) | MN-166 (Early ALS Cohort) (N=34) | Placebo (for MN-166) (Advanced ALS Cohort) (N=8) | MN-166 (Advanced ALS Cohort) (N=11)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (for MN-166) (Early ALS Cohort) (N=17) | MN-166 (Early ALS Cohort) (N=34) | Placebo (for MN-166) (Advanced ALS Cohort) (N=8) | MN-166 (Advanced ALS Cohort) (N=11)
muscle weakness (Musculoskeletal and connective tissue disorders) | 9 (9) | 18 (18) | 1 (1) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 14 (14) | 1 (1) | 5 (5)
Fatigue (General disorders) | 4 (4) | 12 (12) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 9 (9) | 0 (0) | 2 (2)
muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7) | 2 (2) | 3 (3)
nausea (Gastrointestinal disorders) | 2 (2) | 7 (7) | 0 (0) | 0 (0)
weight decreased (Gastrointestinal disorders) | 2 (2) | 7 (7) | 2 (2) | 3 (3)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
injury (Injury, poisoning and procedural complications) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
mobility decreased (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
dysphagia (Gastrointestinal disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
abdominal distention (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
gastrostomy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
edema peripheral (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT02238626/Prot_SAP_000.pdf